CLINICAL TRIAL: NCT00302523
Title: Tacrolimus Treatment of Patients With Idiopathic
Brief Title: Tacrolimus Treatment of Patients With Idiopathic Membranous Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi-Hong Liu, M.D., Research Institute of Nephrology, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0603
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Idiopathic Membranous Nephropathy
Keywords: Idiopathic Membranous Nephropathy; Treatment; Tacrolimus; Cyclophosphamide
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FK506 (Active Comparator)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — FK506,0.1mg/kg/d
  Other Names: Tacrolimus,Prograf

SUMMARY:
The purpose of this study is:

* To explore the potential role of tacrolimus in the treatment of membranous nephropathy.
* To investigate the safety and tolerability of tacrolimus vs methylprednisolone plus cyclophosphamide.

DETAILED DESCRIPTION:
Idiopathic membranous nephropathy is the most common cause of nephrotic syndrome in adults. Over the past decade, a number of studies have reported therapeutic efficacy for treatment with Cyclosporine-A (CSA) in patients with nephrotic syndrome including patients with membranous nephropathy. This study will evaluate the safety and effectiveness of a new calcineurin immunosuppressive drug, tacrolimus (FK506), in reducing the amount of protein in the urine in patients with membranous nephropathy. Forty patients with biopsy-proven membranous nephropathy will be recruited. Candidates must have completed at least six month of treatment with a stable dose of angiotensin converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARBs). They will be screened with a medical history, physical examination, blood tests, and an examination for infection, cancers, and other conditions that can cause membranous nephropathy. The investigators plan to conduct an open-label study of the efficacy and safety of tacrolimus in the treatment of membranous nephropathy. They will be treated with oral tacrolimus for 6 months, followed by 6 months of maintenance. Proteinuria, renal function will be monitored. Complete remission is defined as 24-hour urinary protein excretion to less than 0.4 mg/day. This study will explore the potential role of tacrolimus in the treatment of membranous nephropathy, which is usually resistant to conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven idiopathic membranous nephropathy
* Nephrotic syndrome with proteinuria ( > 4 g/day) and serum albumin < 30 g/dl
* Age 18-60 years with informed consent

Exclusion Criteria:

* Patient with abnormal liver function tests
* Prior therapy with sirolimus, CSA, MMF, or azathioprin, cytoxan, chlorambucil, levamisole, methotrexate, or nitrogen mustard in the last 90 days
* Active/serious infection
* Patient with hepatitis B surface antigen or who is hepatitis C antibody positive
* Patient who is diabetic
* Patient is allergic or intolerant to macrolide antibiotics or tacrolimus

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To explore the potential role of tacrolimus in the treatment of membranous nephropathy. | 18 months

SECONDARY OUTCOMES:
To investigate the safety and tolerability of tacrolimus vs intravenous CTX pulse. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-hong Liu, M.D., Study Director — Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine
Locations (2):
- China (2):
  - Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu
  - Research Institute of Nephrology, Jinling Hospital, Nanjing, Jiangsu

REFERENCES:
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952